CLINICAL TRIAL: NCT04026711
Title: MitoQ for the Treatment of Metabolic Dysfunction in Asthma
Acronym: MIMDA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Anne Dixon, Professor of Medicine, Director of Pulmonary and Critical Care Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0564
Record Dates: First submitted 2019-05-30; First posted 2019-07-19 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity | interventions — mitoquinol; mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double masked study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MitoQ (Active Comparator): MitoQ 40 mg per day for 12 weeks
  Interventions: Drug: Mitoquinol
- Placebo (Placebo Comparator): placebo daily for 12 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Mitoquinol — Mitoquinol (MitoQ) 40 mg per day for 12 weeks
  Other Names: MitoQ
  Arms: MitoQ
Drug: Placebo oral tablet — Placebo daily for 12 weeks
  Arms: Placebo

SUMMARY:
A 14-week, randomized, placebo-controlled, double-masked clinical trial in 40 obese patients with poorly controlled asthma.

The intervention is Mitoquinol (MitoQ) versus placebo.

The primary aim of this pilot study is to determine if MitoQ improves airway reactivity in obese patients with asthma.

DETAILED DESCRIPTION:
Study aim:

The objective of this proposal is to conduct a pilot clinical trial to determine if the mitochondrial-targeted anti-oxidant MitoQ improves airway reactivity in obese patients with poorly controlled asthma.

Type of Study:

A 14 weeks, prospective, two center (Duke and the University of Vermont), randomized, placebo-controlled, double-masked clinical trial.

Study Population:

40 patients with obesity and poorly controlled asthma.

Intervention:

MitoQ 40 mg per day versus placebo.

ELIGIBILITY:
Inclusion criteria:

1. participant reported physician diagnosis of asthma
2. participant reported on regular prescribed controller therapy for at least 3 months
3. positive methacholine challenge (as determined by spirometry PD20 or oscillometry PD50 ≤ 4.0 mg/ml at visit 2)
4. age: ≥18 years
5. BMI ≥ 30 kg/m2 (at visit 1)
6. poorly controlled asthma defined as one of the following:

   1. Asthma Control Test5 Score ≤ 19 (at visit 1), or
   2. Participant reported use of rescue inhaler on average > 2 uses/week for preceding month, or
   3. Participant reported nocturnal asthma awakening on average 1 or more times / week in preceding month, or
   4. Participant reported ED/hospital visit or prednisone course for asthma in past six months
7. ability and willingness to provide informed consent

Exclusion criteria:

1. participant reported use of an investigational agent in the prior 30 days
2. participant reported physician diagnosis of chronic obstructive pulmonary disease
3. pregnancy and/or participant reported lactation
4. females of childbearing age who do not agree to practice an adequate birth control method for the duration of the study (abstinence, combination barrier and spermicide, or hormonal)
5. participant reported greater than 10 pack year smoking history
6. participant reported smoking conventional tobacco products (cigar, cigarette, & pipes) within the last 6 months
7. participant reported e-cigarette use more than 2x/week
8. participant unwilling to withhold e-cigarette use for the duration of the study
9. participant reported vaping more than 2x/week
10. participant unwilling to withhold vaping for the duration of the study
11. participant reported marijuana use (inhalation) more than 2x/week
12. participant unwilling to withhold marijuana use (inhalation) for the duration of the study
13. participant reported sinus surgery performed ≤ 4 weeks from visit 1
14. participant reported eye surgery within the prior 3 months
15. participant reported use of the antioxidants idebenone or co-enzyme Q10 within 8 weeks
16. participant reported tendency to develop severe nose bleeds
17. FEV1 ˂ 60% predicted or < 1.5 Liters at visit 1
18. participant reported treatment for asthma exacerbation in the previous 4 weeks
19. participant was not able to complete at least 50% of the days on the diary cards returned at visit 2
20. other significant disease that in the opinion of the investigator would interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Dixon, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 1/1/2020-12/1/2023 Recruitment locations: two pulmonary clinics at academic medical centers in the U.S.
Pre-assignment Details: Run in period after screening prior to randomization 9 participants excluded 6 screen fails (2 low lung function, 3 negative methacholine, 1 unable to perform study procedures 3 withdrew (1 lack of transport, 2 research burden)
Period: Overall Study
Arm/Group | MitoQ | Placebo
Started | 20 | 18
Completed | 18 | 18
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — mental health crisis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MitoQ | Placebo | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — age in years
  years | 50 (13) | 55 (7) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 18 | 38
Asthma Control Test [Mean (Standard Deviation); unit: total score] — units on scale 5-25, high score indicative of better control
  total score | 16.4 (5.2) | 16.3 (3.1) | 16.3 (4.2)
Marks Asthma Quality of Life [Mean (Standard Deviation); unit: score on questionnaire] — Disease specific quality of life questionnaire: range 1-5, higher score indicative of better quality of life
  score on questionnaire | 2.19 (0.98) | 2.27 (0.76) | 2.23 (0.87)
Airway reactivity to methacholine [Median (Inter-Quartile Range); unit: μg methacholine] — dose of methacholine producing a 20% decrease in FEV1 Population: one participant in the placebo group had poor quality test, and so could not be included in the analysis
  μg methacholine
    number analyzed (Participants) | 20 | 17 | 37
    (all) | 44.5 [6.59 to 441] | 113 [51 to 409] | 110 [44 to 318]
FEV1 [Mean (Standard Deviation); unit: liters] — Forced expiratory volume in 1 second
  liters | 2.45 (0.74) | 2.32 (0.75) | 2.39 (0.74)
FVC [Mean (Standard Deviation); unit: liters] — Forced vital capacity
  liters | 3.48 (1.04) | 3.13 (0.95) | 3.30 (1.03)
AX [Median (Inter-Quartile Range); unit: cm H20/L] — Impedance (Ax, area under the reactance curve)
  cm H20/L | 37.03 [12.76 to 44.21] | 59.06 [35.01 to 73.95] | 42.61 [36.57 to 58.97]

OUTCOME MEASURES:

1. Primary Outcome: Change in Airway Reactivity
Description: change in airway reactivity, measured by change in the concentration of methacholine producing a 20 % decrease in forced expiratory volume in one second, from baseline
Time Frame: Through study completion, 12 weeks
Population: 2 participants in the MitoQ group withdrew 4 participants in the placebo group did not perform methacholine at 12 week visit: Lung function too low (FEV1 less than 60%), and participants unable to complete testing
Measure: Median (Inter-Quartile Range); unit: μg methacholine
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 18 | 14
μg methacholine | 0 [-25.5 to 1.4] | -0.8 [-57 to 0]
Statistical Analysis 1: Comparison: MitoQ vs Placebo; Test type: Superiority; p = 0.81, Wilcoxon rank sum

2. Secondary Outcome: Change in Asthma Control Test (ACT)
Description: To collect data on asthma symptoms measured by asthma control questionnaire with units on a scale from 5-25 (the lower the score, the worse the asthma symptoms)
Time Frame: Through study completion, 12 weeks
Population: 2 withdrew from mitoQ group
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 18 | 18
score | 1 [-1 to 2] | 1 [-2 to 2]

3. Secondary Outcome: Number of Participants With Adherence at 12 Weeks
Description: Adherence determined from pill counts (classified as adherent if used at least 80% of predicted pills)
Time Frame: Through study completion, 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 18 | 18
Participants | 15 | 12

4. Secondary Outcome: Change in Asthma Quality of Life Questionnaire Score
Description: The Marks Asthma Quality of Life Questionnaire (Marks AQLQ). units on a scale from 1 to 5. Higher score indicates better quality of life
Time Frame: Through study completion, 12 weeks
Measure: Median (Inter-Quartile Range); unit: questionnaire score
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 18 | 18
questionnaire score | -0.08 [-0.35 to 0.10] | -0.05 [-0.30 to 0.15]

5. Secondary Outcome: Change in FEV1
Description: Change in forced expiratory volume in one second between baseline and 12 week visit
Time Frame: Through study completion, 12 weeks
Population: one participant unable to complete spirometry testing at 12 week visit
Measure: Median (Inter-Quartile Range); unit: liters
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 18 | 17
liters | -0.01 [0.18 to 0.24] | 0.03 [-0.13 to 0.14]

6. Secondary Outcome: Change in FVC
Description: Change in forced vital capacity from baseline to 12 weeks measured in liters
Time Frame: Through study completion, 12 weeks
Population: one participant in the placebo group unable to perform lung function testing at 12 week visit
Measure: Median (Inter-Quartile Range); unit: liters
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 18 | 17
liters | -0.01 [-0.19 to 0.02] | 0.01 [-0.18 to 0.22]

ADVERSE EVENTS:
Time Frame: From enrollment until study end (after 12 weeks on study drug)
Arm/Group | MitoQ | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 12/20 | 10/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MitoQ (N=20) | Placebo (N=18)
headache (General disorders) | 8 | 6
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 2
gastroesophageal reflux/ nausea (Gastrointestinal disorders) | 7 | 5
diarrhea (Gastrointestinal disorders) | 4 | 5
abdominal pain (Gastrointestinal disorders) | 3 | 3
skin rash (Skin and subcutaneous tissue disorders) | 4 | 2
muscle pain (Musculoskeletal and connective tissue disorders) | 6 | 6
fatigue (General disorders) | 1 | 1
dizziness (General disorders) | 1 | 0
joint pain (Musculoskeletal and connective tissue disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT04026711/Prot_SAP_000.pdf